CLINICAL TRIAL: NCT06132568
Title: VITALYST EFS: VITALYST Temporary Percutaneous Transvalvular Circulatory Support System Early Feasibility Study
Brief Title: VITALYST Early Feasibility Study in High-Risk PCI Patients (VITALYST EFS)
Acronym: VITALYST EFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: S2496
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: High-risk Percutaneous Coronary Intervention; Heart Disease, Coronary
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- High Risk PCI Patients (Experimental): Patients undergoing non-emergent, high-risk percutaneous coronary interventions
  Interventions: Device: VITALYST System

INTERVENTIONS:
Device: VITALYST System — The VITALYST System is a temporary ventricular support device indicated for use during high-risk percutaneous coronary interventions (HR-PCI) performed electively in hemodynamically stable subjects with severe coronary artery disease.
  Other Names: Percutaneous Mechanical Circulatory Support

SUMMARY:
The VITALYST Early Feasibility study (EFS) is designed to evaluate the feasibility and safety of the VITALYST System in subjects undergoing elective high-risk percutaneous coronary intervention (HR-PCI).

DETAILED DESCRIPTION:
The VITALYST EFS is a prospective, open-label, single-arm, multicenter feasibility study of the VITALYST System.

The VITALYST System will be used to provide temporary circulatory support in patients undergoing non-emergent high risk percutaneous interventions (HR-PCI).

ELIGIBILITY:
Inclusion Criteria:

* Subject provides signed informed consent.
* Subject is ≥ 18 years and < 90 years of age.
* Subject is indicated for NON-emergent PCI of at least one de novo or restenotic lesion in a native coronary vessel or coronary artery bypass graft (CABG) and has left ventricular ejection fraction (LVEF) ≤ 50% with the following: Unprotected left main or Last remaining vessel or Three vessel disease (at least one ≥ 50% diameter stenosis based on center's visual assessment in all three major epicardial territories)
* Heart team, which must include a cardiac surgeon, agrees that HR-PCI is appropriate.

Exclusion Criteria:

* Subject has had STEMI within 72 hours with persistent elevation of cardiac enzymes.
* Subject has had pre-procedure cardiac arrest requiring CPR within 24 hours of enrollment.
* Subject has systolic blood pressure < 90 mmHg with evidence of end organ hypoperfusion (e.g., cool extremities or urine < 30 mL/hour).
* Subject has had need for inotropes/vasopressors or mechanical circulatory support (including intra-aortic balloon pump) in the previous 24 hours to maintain a systolic blood pressure ≥ 90 mmHg.
* Subject has left ventricular mural thrombus.
* Subject has a prosthetic aortic valve.
* Subject has pericarditis or constrictive heart disease (constrictive pericarditis or restrictive cardiomyopathy).
* Subject has moderate or greater aortic valve stenosis or moderate or greater aortic valve insufficiency (by echocardiographic assessment, graded as > 2+).
* Subject has abnormalities of the aorta that preclude safe delivery of the device, including severe calcification, tortuosity, aneurysm, or prior surgery.
* Subject has PVD preventing passage of the device (e.g., calcification, small caliber) or tortuosity that would preclude safe placement of the introducer sheath as per the IFU.
* Subject is not on dialysis and has creatinine > 4 mg/dL.
* Subject has a history of liver dysfunction (Childs Class C) with elevation of liver enzymes and bilirubin > 3× ULN or INR ≥ 2.
* Subject has had a recent (within 30 days) stroke or TIA.
* Subject has known hypersensitivity to intravenous contrast agents that cannot be adequately pre-medicated or has known hypersensitivity to heparin, aspirin, ADP receptor inhibitors or nitinol.
* Subject has current or a history of heparin induced thrombocytopenia.
* Subject has uncorrected abnormal coagulation or platelet count ≤ 75,000/mm³ or INR ≥ 2.0.
* Subject has significant right heart failure based on any one of the following criteria: RVSWI < 0.30 mmHg·L/m² or PVR > 3.6 Woods units or Pulmonary artery pulsatility index < 1.85
* Subject requires non-elective mechanical ventilation.
* Subject has an atrial or ventricular septal defect (including post-infarct VSD).
* Subject has left ventricular rupture.
* Subject has cardiac tamponade.
* Subject has severe pulmonary disease (FEV1 < 1L).
* Subject has sustained or non-sustained ventricular tachycardia.
* Subject is breast feeding or is pregnant.
* Subject has infection of the proposed procedural access site or active systemic infection.
* Subject has any condition that requires premature discontinuation of recommended antiplatelet and/or anticoagulant therapy before 90 days following the index procedure.
* Any use of a mechanical circulatory support device within 14 days prior to the index procedure.
* Staged PCI is planned within 90 days following device removal.
* Subject is participating in another investigational drug or device study that has not reached its primary endpoint.
* Subject has other disease condition(s) resulting in the subject being unsuitable for participation in the clinical trial (e.g., advanced malignancy with limited expected survival)
* Subject has other disease condition(s) which the Investigator has determined may cause non-compliance to the study requirements.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Clinical Success | Measured through 72 hours or hospital discharge (whichever comes first) after the intervention/procedure
  The primary endpoint consists of the composite endpoint of Clinical Success [measured through 72 hours or hospital discharge (whichever comes first)], which is defined as follows.
  * Technical Success: Successful delivery of the device to the correct anatomical position; and Successful operation and removal of the VITALYST circulatory support system
  * Absence of termination of revascularization procedure due to hemodynamic concern, or escalation to ECMO or other more intensive mechanical circulatory support device, or the use of vasopressors or inotropes
  * No conversion to open heart surgery
  * No mortality

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Piedmont Heart Institute, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
- Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html)